CLINICAL TRIAL: NCT00333684
Title: A Prospective Study Evaluating the Safety, Efficacy and Psychological Effects of Treating Antiretroviral Drug-Induced Facial Lipoatrophy With Bio-Alcamid Soft Tissue Endoprosthesis
Brief Title: Safety, Efficacy and Psychological Effects of Treating Antiretroviral Drug-Induced Facial Lipoatrophy With Bio-Alcamid
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Immunodeficiency Research Collaborative (Other)
Collaborators: Pur Medical Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LA-BA-001
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Human Immunodeficiency Virus; Facial Lipoatrophy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

ARMS (2):
- receive bioalcamid at baseline (Active Comparator): half subjects received bioalcamid at baseline
  Interventions: Device: BIO-ALCAMID SOFT TISSUE ENDOPROSTHESIS
- Receive bioalcamid at 24 weeks (Active Comparator): other half of subjets received bioalcamid at 24 weeks
  Interventions: Device: BIO-ALCAMID SOFT TISSUE ENDOPROSTHESIS

INTERVENTIONS:
Device: BIO-ALCAMID SOFT TISSUE ENDOPROSTHESIS — prosthetic bioalcamid was injected- amounts determined by the plastic surgeon and depended individual needs

SUMMARY:
Evaluate and record any changes in the Quality of Life and psychological state of the affected study group following treatment with Bio-Alcamid.

Evaluate the safety and efficacy of Bio-Alcamid for restoring the natural fullness and contours of the face affected by HIV drug-induced lipoatrophy. Pre-treatment classification and post treatment recording of changes will be performed by, both, the Principal Investigator and the Treatment Specialist and independently by a 'Blinded' Co-Investigator at post treatment Week 12.

Safety data for Bio-Alcamid will be collected throughout the duration of the study. Safety will be determined by the rates of procedure-related events and adverse experiences associated with the use of Bio-Alcamid.

DETAILED DESCRIPTION:
Thirty (30) participants in the randomized portion of the study will be selected who have been classified as having moderate to severe facial lipoatrophy based on the three investigators evaluations.

These patients will be divided into two groups -

The Treatment Group - 15: At Day -1, the Treatment group will be established by the inclusion/exclusion criteria and consent forms will be signed. At Day 0 they will complete QOL Surveys and will receive treatment with Bio-Alcamid in the affected facial area(s). At Day 7, they will return to complete the QOL Surveys and allow the CITS to determine if a touch-up is necessary. If so, one touch-up session is permitted at week 6. The participants will again complete QOL Surveys and have efficacy assessments at week 12. The Treatment Group will continue with follow-up sessions at week 24, 48, 60 and at 96 weeks. Professional clinical photographs will be taken at each visit.

The Control Group - 15: At Day -1, the Control group will be established by the inclusion/exclusion criteria and consent forms will be signed. At Day 0, they will complete QOL Surveys. They will return for visits at baseline and week 6 as well to complete QOL Surveys. At Week 12, they will complete the QOL Surveys and will receive a BA treatment. At Week 13, they will return to complete the QOL Surveys and allow the CITS to determine if a touch-up is necessary. If so, one touch-up session is permitted at week 18. If not, these participants will again complete QOL Surveys and have efficacy assessments at week 24. The Control Group will continue with follow-up sessions at week 48, 60, 96 and at 104 weeks. Professional clinical photographs will be taken at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Have moderate to severe levels of facial lipoatrophy determined by the three investigstors
* If female of child-bearing potential (not menopausal for at least 1 year nor surgically sterile), have a negative urine pregnancy test prior to any study treatments and be willing to use oral contraception or another medically acceptable form of contraception for the duration of the study
* Be able to understand and comply with the requirements of this study
* Be willing and able to provide written Informed Consent prior to any study-related procedures being performed
* Agree to refrain from seeking other treatment for lipoatrophy in the facial area while participating in this study

Exclusion Criteria:

* Are pregnant, lactating, or trying to become pregnant
* Had prior therapy (e.g., other permanent or biodegradable injectable fillers or surgical correction such as a face-lift, etc.) within 9 months prior to entry into the study or are planning to undergo such therapy during the study
* Have any active inflammation, infection, or unhealed wound of the face
* Have any contraindicated condition described in the package insert for the product to be administered.
* Have a history of anaphylaxis or multiple severe allergies.
* Have planned relocation during the study, which would make follow-up visits impossible during the course of the study
* Used aspirin or nonsteroidal anti-inflammatory drugs (NSAIDs) within 1 week prior to initial or touch-up treatment or are taking concomitant anticoagulant therapy, anti-platelet therapy, or have a history of bleeding disorders
* Used over-the-counter wrinkle products (e.g., alpha-hydroxy acids) or prescription treatments (e.g., Renova, Retin-A, microdermabrasion, chemical peels) in the facial area within 4 weeks prior to study start. In addition, participants will be restricted from using over-the-counter wrinkle products or prescription treatments to the facial area for the duration of the study.
* Have received any investigational product within 30 days prior to study enrollment or are planning to receive other investigational products during the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2004-12; Primary Completion 2006-11 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To evaluate Quality of Life using the slightly modified Dermatology Quality Life Survey and the MOS-HIV Survey. | 96 weeks
  To evaluate Quality of Life using the slightly modified Dermatology Quality Life Survey and the MOS-HIV Survey.

SECONDARY OUTCOMES:
Evaluate the safety and efficacy of Bioalcamid for restoring the natural fullness and contours of the face affected by HIV drug-induced lipoatrophy. | 96 weeks
  valuate the safety and efficacy of Bioalcamid for restoring the natural fullness and contours of the face affected by HIV drug-induced lipoatrophy.

CONTACTS AND LOCATIONS:
Overall Officials: Mona Loutfy, MD, FRCP(C), Principal Investigator — Canadian Immunodeficiency Research Collaborative
Locations (1):
- Maple Leaf Medical Clinic, Toronto, Ontario, Canada